CLINICAL TRIAL: NCT02839954
Title: Study Evaluating the Efficacy and Safety of Chimeric Antigen Receptor-Modified pNK Cells in MUC1 Positive Advanced Refractory or Relapsed Solid Tumor
Brief Title: CAR-pNK Cell Immunotherapy in MUC1 Positive Relapsed or Refractory Solid Tumor
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Collaborators: The First People's Hospital of Hefei (Other); Hefei Binhu Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-121-001
Record Dates: First submitted 2016-07-14; First posted 2016-07-21 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Hepatocellular Carcinoma; Non-small Cell Lung Cancer; Pancreatic Carcinoma; Triple-Negative Invasive Breast Carcinoma; Malignant Glioma of Brain; Colorectal Carcinoma; Gastric Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms; Colorectal Neoplasms; Stomach Neoplasms | interventions — Sensitivity and Specificity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CAR-pNK Cell immunotherapy (Experimental): Enrolled patients will receive CAR-pNK cell immunotherapy with a novel specific chimeric antigen receptor targeting MUC1 antigen by infusion.
  Interventions: Biological: anti-MUC1 CAR-pNK cells

INTERVENTIONS:
Biological: anti-MUC1 CAR-pNK cells
  Other Names: Chimeric antigen receptor NK cells with specificity for MUC1

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of CAR-pNK cell immunotherapy in patients with MUC1 positive relapsed or refractory solid tumor.

ELIGIBILITY:
Inclusion Criteria:

Male and female subjects with MUC1+ malignancies in patients with no available curative treatment options who have limited prognosis (several months to < 2 year survival) with currently available therapies will be enrolled:

1. Eligible diseases: MUC1+ malignant glioma of brain, colorectal carcinoma, gastric carcinoma, hepatocellular carcinoma, non-small cell lung cancer, pancreatic carcinoma and triple-negative basal-like breast carcinoma.
2. Patients 18 years of age or older, and must have a life expectancy > 12 weeks.
3. MUC1 is expressed in malignancy tissues by immuno-histochemical (IHC).
4. Eastern cooperative oncology group (ECOG) performance status of 0-2 or karnofsky performance status (KPS) score is higher than 60.
5. Presence of measurable disease by RECIST.
6. Females of child-bearing potential must have a negative pregnancy test and all subjects must agree to use an effective method of contraception for up to two weeks after the last infusion of CAR-pNK cells.
7. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements: White blood cell count (WBC) ≥ 2500c/ml, Platelets ≥ 50×10^9/L, Hb ≥ 9.0g/dL, lymphocyte (LY) ≥ 0.7×10^9/L, LY% ≥ 15%, Alb ≥ 2.8g/dL, serum lipase and amylase < 1.5×upper limit of normal, serum creatinine ≤ 2.5mg/dL, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5×upper limit of normal, serum total bilirubin ≤ 2.0mg/dL. These tests must be conducted within 7 days prior to registration.
8. Ability to give informed consent.

Exclusion Criteria:

1. Patients with symptomatic central nervous system (CNS) involvement.
2. Pregnant or nursing women may not participate.
3. Active HIV, hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
4. Serious illness or medical condition which would not permit the patient to be managed according to the protocol, including active uncontrolled infection, major cardiovascular, coagulation disorders, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive/restrictive pulmonary disease, or psychiatric or emotional disorders.
5. Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary.
6. The existence of unstable or active ulcers or gastrointestinal bleeding.
7. Patients with a history of organ transplantation or are waiting for organ transplantation.
8. Patients need anticoagulant therapy (such as warfarin or heparin).
9. Patients need long-term antiplatelet therapy (aspirin at a dose > 300mg/d; clopidogrel at a dose > 75mg/d).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Phase I: Adverse events attributed to the administration of the anti-MUC1 CAR-pNK cells | 2 years
  Determine the toxicity profile of the MUC1 targeted CAR-pNK cells with Common Toxicity Criteria for Adverse Effects (CTCAE) version 4.0.

SECONDARY OUTCOMES:
Phase II: Objective Response Rate | 2 years
  The objective response rate (ORR) is defined as the proportion of patients who achieve radiographic partial or complete response (PR or CR) according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 guideline.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Yang, Ph.D., Principal Investigator — PersonGen BioTherapeutics (Suzhou) Co., Ltd.
Locations (1):
- PersonGen BioTherapeutics (Suzhou) Co., Ltd., Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Del Zotto G, Marcenaro E, Vacca P, Sivori S, Pende D, Della Chiesa M, Moretta F, Ingegnere T, Mingari MC, Moretta A, Moretta L. Markers and function of human NK cells in normal and pathological conditions. Cytometry B Clin Cytom. 2017 Mar;92(2):100-114. doi: 10.1002/cyto.b.21508. Epub 2017 Feb 12. PMID 28054442